CLINICAL TRIAL: NCT00397722
Title: Study CRH103390: A 12 Week Flexible Dose Study of GW876008, Placebo and Active Control (Paroxetine) in the Treatment of Social Anxiety Disorder (SocAD)
Brief Title: Treatment Of Patients With Social Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CRH103390
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Social Phobia
Keywords: safety; outpatients with a diagnosis of Social Anxiety disorder (SocAD).; effectiveness
MeSH Terms: conditions — Phobia, Social | interventions — GW 876008; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW876008
Drug: paroxetine
  Other Names: GW876008

SUMMARY:
GW876008 is a drug which may change mans reaction to stress, by decreasing the fear, physical and behavior symptoms that people with SocAD experience in social situations.

ELIGIBILITY:
Inclusion criteria:

* are diagnosed with generalized social anxiety disorder/social phobia.

Exclusion criteria:

* have a diagnosis of major depressive disorder
* have a history of Schizophrenia, Schizoaffective Disorder, or Bipolar Disorder.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 299 (Actual)
Dates: Start 2006-11-09 (Actual); Primary Completion 2007-09-05 (Actual); Study Completion 2007-09-05 (Actual)

PRIMARY OUTCOMES:
Change from randomization in the clinician-administered LSAS total score at the end of the treatment phase (Week 12) | Baseline (Day 0) and Week 12
  The LSAS is an investigator-rated scale consisting of 48 questions concerning various social situations. The LSAS is the first psychiatric assessment at all post-screening visits. A qualified independent efficacy rater scored the participant's "fear or anxiety" and "avoidance" of social situations on 4-point scale : where, 0= None, 1= Mild, 2= Moderate, 3= Severe. Scores were recorded in participant's source documents. The LSAS total score was the sum of each of the forty-eight individual responses. Day 0 was Baseline and change from Baseline was calculated by subtracting Baseline value from Week 12 value. Data for adjusted mean and SE is presented.
Change from randomization on the LSAS Fear subscale score at Week 12 | Baseline (Day 0) Week 12
  The LSAS consisted of 24 fear responses. All individual items were rated on a scale 0 (none) -3 (severe) with higher scores indicating more severe fear. The LSAS fear subscale score was the sum of each of the 24 individual responses. If at least 22 items of the items making up the subscale of interest were present at a particular time point, the subscale score was calculated as Sum of non-missing items multiplied with 24/Number of non-missing items. If less than 22 of the items making up the score of interest were available for a participant at a particular time point, the subscale score was not calculated for that time point. Day 0 was Baseline and change from Baseline was calculated by subtracting Baseline value from Week 12 value. Data for adjusted mean and SE is presented.
Change from randomization on the LSAS Avoidance subscale score at Week 12 | Baseline (Day 0) and Week 12
  The LSAS consisted of 24 avoidance responses. All individual items were rated on a scale 0 (never) -3 (always) with higher scores indicating more severe avoidance. The LSAS avoidance subscale Score was the sum of each of the 24 individual responses. If at least 22 items of the items making up the subscale of interest were present at a particular time point, the total score was calculated as Sum of non-missing items multiplied with 24/Number of non-missing items. If less than 22 of the items making up the score of interest were available for a participant at a particular time point, the subscale score was not calculated for that time point. . Day 0 was Baseline and change from Baseline was calculated by subtracting Baseline value from Week 12 value. Data for adjusted mean and SE is presented.
Change from randomization on the Social Avoidance and Distress Scale (SADS) total score at Week 12 | Baseline (Day 0) and Week 12
  The SADS is a 28 item questionnaire. The total score was obtained by summing together the responses for all 28 items from the SADS questionnaire. Each individual item was rated as true or false. One point was given where items 2, 5, 8, 10, 11, 13, 14, 16, 18, 20, 21, 23, 24, 26 were marked as true and 1 point when each of the remaining items were marked as false. This gave a possible range of possible scores from 0 to 28 with higher scores indicating more severe disorder. If at least 26 of the items making up the total score were present at a particular time point, the total score was calculated as Sum of scores for non-missing items multiplied with 28/Number of non-missing items. If less than 26 of the items making up the score of interest were available for a participant at a particular time point, the total score was not calculated for that time point.

SECONDARY OUTCOMES:
Number of participants with abnormal electrocardiogram (ECG) findings any time post randomization | Up to Week 12
  All 12-lead ECGs were digitally acquired by a qualified clinician and transmitted to a specified central laboratory. The ECG traces were interpreted by a qualified physician. Number of participants with abnormal ECG findings were reported.
Change from Randomization in Vital Signs: systolic and diastolic blood pressure (SBP and DBP) | Baseline (Day 0) Up to Week 12
  Vital signs were measured at all scheduled study visits which included SBP and DBP. Change from Baseline values were presented for SBP and DBP. Day 0 was Baseline and change from Baseline was calculated by subtracting Baseline value from value at scheduled study visits. Data presented for maximum (max) increase-decrease in SBP/DBP.
Change from Randomization in vital signs : heart rate | Baseline (Day 0) and up to Week 12
  Vital signs were measured at all scheduled study visits which included heart rate. Change from Baseline values were presented for heart rate. Day 0 was Baseline and change from Baseline was calculated by subtracting Baseline value from value at scheduled study visits. Data presented for max increase-decrease in heart rate.
Number of participants with chemistry data outside the normal range (Any time post-Randomization) | Up to Week 12
  Number of participants with chemistry values outside the normal range up to 12 weeks were presented. Chemistry parameters included: Calcium, Bicarbonate, Chloride, Creatine Kinase, Creatinine, Magnesium, Phosphorus, Potassium, Sodium, Urea and Uric Acid.
Number of participants with hematology data outside the normal range (Any time post-Randomization) | Up to Week 12
  Number of participants with hematology values outside the normal range up to 12 weeks were presented. Hematology parameters included: Basophils, Eosinophils, Hematocrit, Hemoglobin, Lymphocytes, Mean Corpuscular Hemoglobin (MCH), Mean Corpuscular Hemoglobin Concentration (MCHC), Mean Corpuscular Volume (MCV), Monocytes, Platelet count, Red blood cell, Total neutrophils and White blood cells.
Number of participants with All adverse events (AE) and serious adverse events SAE) | Up to 18 Weeks
  Data for number of participants who presented one or more adverse events (serious or non serious) was reported. An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Trough Concentration (Ctrough) | Up to Week 12 (pre dose)
  Ctrough is the lowest concentration reached by a drug before the next dose is administered. Blood samples for Pharmacokinetic assessment were collected pre dose at Week 1, Week 2, Week 4, Week 8 and Week 12.
Exposure at steady state (AUC (0-τ)) | Up to Week 12
  Blood samples for Pharmacokinetic assessment were collected pre dose at Week 1, Week 2, Week 4, Week 8 and Week 12. for AUC (0-τ)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- United States (12):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Temecula, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Smyrna, Georgia
  - GSK Investigational Site, Oakbrook Terrace, Illinois
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Farmington Hills, Michigan
  - GSK Investigational Site, Nutley, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Media, Pennsylvania
- Canada (4):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Miramichi, New Brunswick
  - GSK Investigational Site, Mississauga, Ontario
- Finland (3):
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Rauma
  - GSK Investigational Site, Turku
- Germany (5):
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Westerstede, Lower Saxony
  - GSK Investigational Site, Berlin
- Norway (3):
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Sandvika
- South Africa (3):
  - GSK Investigational Site, Tygerberg, Eastern Cape
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Observatory ,Cape Town
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Uppsala